CLINICAL TRIAL: NCT01006187
Title: Comparison of Different Analgesic Methods for Reducing Pain From Adult Intramuscular Influenza Virus Vaccine Injection
Brief Title: Comparison of Different Methods for Reducing Pain From Influenza Vaccine Injections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Dr. Anna Taddio, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000014280
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Pain; Anxiety
Keywords: Analgesics; Influenza; Vapocoolant; vaccination; pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Influenza, Human | interventions — Maxilene; Osteogenesis, Distraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): 1 liposomal lidocaine 4% cream .
  Interventions: Drug: Liposomal lidocaine
- Group 2 (Active Comparator): Vapocoolant spray
  Interventions: Drug: Vapocoolant spray
- Group 3 (Active Comparator): Rubbing adjacent to the injection site
  Interventions: Other: Rubbing adjacent to the injection site
- Group 4 (Active Comparator): Distraction by means of self-selected reading material or internet
  Interventions: Other: Distraction

INTERVENTIONS:
Drug: Liposomal lidocaine — 4% cream; approximately one gram applied to injection site under an occlusive dressing for 20 minutes prior to injection
  Other Names: Maxilene™
  Arms: Group 1
Drug: Vapocoolant spray — medium stream spray on arm for 4-10 seconds prior to injection
  Other Names: PainEase™
  Arms: Group 2
Other: Rubbing adjacent to the injection site — rubbing adjacent to the injection site before and during injection
  Arms: Group 3
Other: Distraction — By means of self-selected reading material or video
  Arms: Group 4

SUMMARY:
The purpose of this study is to compare four different analgesic strategies in adults undergoing routine influenza immunization

DETAILED DESCRIPTION:
In this study, we will compare relative effectiveness of 4 analgesic strategies (i.e., topical local anesthetics, vapocoolant spray, tactile stimulation and distraction) in adults undergoing routine immunization in order to provide further evidence of the effectiveness of each intervention and to determine if one method is superior to another. We are not including a 'no treatment' group because we do not wish to subject participants to unnecessary pain when there are available analgesic treatments. Moreover, in the presence of a 'no treatment' group, we cannot rule out a placebo effect for all treatment groups unless we provide a matched placebo for each intervention, which is not feasible. In future studies, we plan to address the added benefit of combining analgesic interventions (i.e., evaluating the effect of a multimodal approach).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged >18 years of age undergoing voluntary immunization with influenza virus vaccine

Exclusion Criteria:

* Pre-medication with any of the analgesic interventions in this study,
* Chronic pain syndromes/conditions
* Receiving systemic analgesics and sedatives
* Abnormal circulation (e.g., Raynaud's phenomenon)
* Allergy/hypersensitivity to amide local anesthetics
* Allergy to influenza virus vaccine or constituents
* Prior participation in the trial
* Inability to understand the VAS
* If suspected to be pregnant, pregnant or breastfeeding (due to possible treatment with liposomal lidocaine).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pain from adult intramuscular influenza virus injection | 1 day

SECONDARY OUTCOMES:
Adverse Events | 1 day
Anxiety | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Taddio A, Lord A, Hogan ME, Kikuta A, Yiu A, Darra E, Bruinse B, Keogh T, Stephens D. A randomized controlled trial of analgesia during vaccination in adults. Vaccine. 2010 Jul 19;28(32):5365-9. doi: 10.1016/j.vaccine.2010.05.015. Epub 2010 May 16. PMID 20483194